CLINICAL TRIAL: NCT07079865
Title: Effect of 60-day Peripheral Nerve Stimulation (PNS) in Alleviating Pain and Improving Function After Acute Thoracolumbar Compression Fracture
Status: Recruiting | Type: Observational
Sponsor: Saint Peters University Hospital (Other)
Collaborators: University Orthopaedic Associates (Unknown)
Responsible Party: Sponsor
Other Study IDs: IRB-FY2024-41
Record Dates: First submitted 2025-07-07; First posted 2025-07-23 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-08

CONDITIONS: Thoracolumbar Compression Fractures

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: SPRINT PNS modulation system — Participants will receive treatment using the commercially available SPRINT PNS system. Their pain levels will be assessed using qualified scales including NRS and BPI and their quality of life using the PROMIS scale.

SUMMARY:
The purpose of this study is to track and investigate the outcomes of female patients with acute thoracolumbar compression fractures, focusing on pain management and functional improvement. The study will investigate patients whose compression fractures are within 3 months or less and measure pain scores, using the Numeric Rating Scale (NRS) and Brief Pain Inventory (BPI) and quality of life using the PROMIS questionnaire at 1-week prior to intervention and then 2 weeks, 3 months and 6 months post PNS implantation.

The primary aim is to assess pain reduction among participants that receive the 60-day PNS intervention. The secondary aim is to analyze functional outcomes and quality of life documented in PROMs (Patient Reported Outcomes Measures) provided by CareSense a digital data collection system.

ELIGIBILITY:
Inclusion Criteria:

* Adult females ages 18+
* Osteoporosis diagnosis with acute/subacute insufficiency fractures of the thoracic or lumbar spine identified on MRI or X-ray with significant pain and activity limitation.
* Onset of pain from associated fracture should be less than 3 months.
* Minimum pain should be 4 or greater (Moderate) on the NRS scale and/or impairing their daily activity.
* Patients reported pain should be despite OTC medication trials of NSAIDs, Tylenol, lidocaine patches or similar medications.
* Patients may be taking opioids while receiving treatment however as per routine practice, no additional opioids will be prescribed during the PNS intervention.

Exclusion Criteria:

* Patients with pathological fractures, other etiologies of fracture such as pagets disease, multiple myeloma, local or systemic infection, untreated coagulopathy, untreated psychosocial disease.
* Other etiologies of osteoporosis other than primary osteoporosis will be excluded such as hyperparathyroidism, anorexia, malabsorption, hyperthyroidism, or overtreatment of hypothyroidism, chronic renal failure, cushing.
* Patients with diminished mental capacity (mental condition that will inhibit their ability to complete the assessments) as determined by the investigator.
* Patients with an active cardiac implant device such as a pacemaker or defibrillator.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatient Orthopedic Clinic
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2025-08-07 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in Pain | Baseline (pre-SPRINT PNS) to 2 Weeks Post, 3 Months Post and 6 Months Post Implantation
  Pain as measured using a numeric rating scale (NRS). A 0 - 10 point scale with 0 representing no pain, 1-3 mild, 4-6 moderate and 7-10 severe.
Change in Pain | Baseline (pre-SPRINT PNS) to 2 Weeks Post, 3 Months Post and 6 Months Post Implantation
  Pain as measured using a Brief Pain Inventory (BPI). A 0 - 10 point scale with 0 representing no pain and 10 representing severe pain.

SECONDARY OUTCOMES:
Change in Quality of Life (QOL) | Baseline (pre-SPRINT PNS) to 2 Weeks Post, 3 Months Post and 6 Months Post Implantation
  QOL as measured by PROMIS (Patient-Reported Outcomes Measurement Information System). Responses are scored on 20 to 80 point scale. Scores between 20-55 are within normal limits. Scores 55+ will fall within mild-moderate-severe.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University Orthopaedic Associates, Avenel, New Jersey
  - University Orthopaedic Associates, Morganville, New Jersey
  - University Orthopaedic Associates, Somerset, New Jersey

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Johnell O, Kanis J. Epidemiology of osteoporotic fractures. Osteoporos Int. 2005 Mar;16 Suppl 2:S3-7. doi: 10.1007/s00198-004-1702-6. Epub 2004 Sep 8. PMID 15365697
- [Background] Gautam S, Gopal VG, Khuba S, Agarwal A, V M, Kumar S. Evaluation of the role of vertebral augmentation in chronic vertebral compression fractures: A retrospective study. Interv Pain Med. 2023 Mar 11;2(1):100242. doi: 10.1016/j.inpm.2023.100242. eCollection 2023 Mar. PMID 39239614
- [Background] Chitneni A, Berger AA, Orhurhu V, Kaye AD, Hasoon J. Peripheral Nerve Stimulation of the Saphenous and Superior Lateral Genicular Nerves for Chronic Pain After Knee Surgery. Orthop Rev (Pavia). 2021 May 31;13(2):24435. doi: 10.52965/001c.24435. eCollection 2021. PMID 34745463
- [Background] Huntoon MA, Slavin KV, Hagedorn JM, Crosby ND, Boggs JW. A Retrospective Review of Real-world Outcomes Following 60-day Peripheral Nerve Stimulation for the Treatment of Chronic Pain. Pain Physician. 2023 May;26(3):273-281. PMID 37192232
- [Background] Gabriel RA, Ilfeld BM. Acute postoperative pain management with percutaneous peripheral nerve stimulation: the SPRINT neuromodulation system. Expert Rev Med Devices. 2021 Feb;18(2):145-150. doi: 10.1080/17434440.2021.1877134. Epub 2021 Jan 20. PMID 33446005
- [Background] Buchbinder R, Johnston RV, Rischin KJ, Homik J, Jones CA, Golmohammadi K, Kallmes DF. Percutaneous vertebroplasty for osteoporotic vertebral compression fracture. Cochrane Database Syst Rev. 2018 Apr 4;4(4):CD006349. doi: 10.1002/14651858.CD006349.pub3. PMID 29618171
- [Background] Bernhard J, Heini PF, Villiger PM. Asymptomatic diffuse pulmonary embolism caused by acrylic cement: an unusual complication of percutaneous vertebroplasty. Ann Rheum Dis. 2003 Jan;62(1):85-6. doi: 10.1136/ard.62.1.85. No abstract available. PMID 12480681
- [Background] Prince RL, Lewis JR, Lim WH, Wong G, Wilson KE, Khoo BC, Zhu K, Kiel DP, Schousboe JT. Adding Lateral Spine Imaging for Vertebral Fractures to Densitometric Screening: Improving Ascertainment of Patients at High Risk of Incident Osteoporotic Fractures. J Bone Miner Res. 2019 Feb;34(2):282-289. doi: 10.1002/jbmr.3595. Epub 2018 Nov 5. PMID 30395687
- [Background] Wright NC, Looker AC, Saag KG, Curtis JR, Delzell ES, Randall S, Dawson-Hughes B. The recent prevalence of osteoporosis and low bone mass in the United States based on bone mineral density at the femoral neck or lumbar spine. J Bone Miner Res. 2014 Nov;29(11):2520-6. doi: 10.1002/jbmr.2269. PMID 24771492